CLINICAL TRIAL: NCT00173914
Title: The Association of Endothelial Dysfunction and Cardiac Allograft Vasculopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9200000478; NTUH 92M011
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Heart Transplantation
Keywords: 1. Transplant vasculopathy; 2. Endothelial dysfunction; 3. Myocardial perfusion imaging; 4. Intravascular vascular ultrasound

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Progressive cardiac allograft vasculopathy (CAV) is a serious complication in long-term survivors after heart transplantation. Therefore, we hypothesize that CAV is a diffuse and progressive process, and endothelial function may play an important role in predicting clinical outcome after heart transplantation. Therefore, this single-blinded study is designed to evaluate endothelial function, microvascular flow response and morphology of coronary artery in cardiac allografts,

1. The simultaneous use of IVUS and Doppler wire instrumentation in different pharmacological stress;
2. Tl-201 SPECT (dipyridamole stress/rest); to evaluate the correlation of endothelial function, coronary morphology change and Tl-201 dipyridamole stress myocardial perfusion image.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant receipients who undergoing the coronary angiographic follow-up as standard protocols.

Exclusion Criteria:

1. Acute illness conditions including infection, congestive heart failure (NYHA Fc III, IV), etc.
2. Coronary angiographic finding: coronary stenosis>30% (as grade III, IV by Klauss V et al, Am J Cardiol 1995; 76:463-6).
3. Creatinine >3.0 mg/dl

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Ming Lee, MD, phD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan